CLINICAL TRIAL: NCT00297453
Title: Smoking Treatment in HIV Clinical Care Settings
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Gary Humfleet, Associate Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA 09253-7; P50DA009253 (NIH)
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Internet (Experimental): Individual counseling + nicotine replacement. 6 sessions across a 3 month period.
  Interventions: Behavioral: Internet-based smoking treatment
- Counseling (Experimental): Individual counseling plus nicotine replacement treatment.
  Interventions: Behavioral: Individual Counseling
- Self-Help (Active Comparator): Self-help Manual plus nicotine replacment treatment.
  Interventions: Behavioral: self-help

INTERVENTIONS:
Behavioral: Internet-based smoking treatment — All participants have access to an Internet-based self-help intervention that includes social support through message boards. All participants have access to 10 weeks of nicotine replacement treatment.
  Arms: Internet
Behavioral: Individual Counseling — Six individual counseling sessions are provided over a 12 week treatment period. Participants also have access to a 10-week nicotine replacement treatment.
  Arms: Counseling
Behavioral: self-help — Participants receive a self-help manual and have access to a 10 nicotine replacement treatment.
  Arms: Self-Help

SUMMARY:
The study is designed to evaluate and compare the efficacy and cost effectiveness of 3 smoking cessation treatments with HIV-positive cigarette smokers. The treatments include face-to-face individual counseling, a computer-Internet-based self-help treatment and a self-help manual treatment.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* 18 years or older
* smoking "most days" during the past month
* must be able to read English

Exclusion Criteria:

* any contraindications for over-the-counter nicotine replacement treatment
* active psychotic symptoms
* severe cognitive deficits/dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2006-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
7 day point prevalence biochemically verified abstinence rates | 3, 6, 9, and 12 months following treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Gary Humfleet, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Mdege ND, Shah S, Dogar O, Pool ER, Weatherburn P, Siddiqi K, Zyambo C, Livingstone-Banks J. Interventions for tobacco use cessation in people living with HIV. Cochrane Database Syst Rev. 2024 Aug 5;8(8):CD011120. doi: 10.1002/14651858.CD011120.pub3. PMID 39101506